CLINICAL TRIAL: NCT01083550
Title: Decision Aid on Radioactive Iodine Treatment for Early Stage Papillary Thyroid Cancer (Randomized Controlled Trial)
Brief Title: Decision Making on Radioactive Iodine Treatment for Papillary Thyroid Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REB 09-0986-BE; UHNREB 09-0986-BE (Other: University Health Network Research Ethics Board Number)
Record Dates: First submitted 2010-02-24; First posted 2010-03-09 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Thyroid Cancer
Keywords: thyroid carcinoma; thyroid cancer; therapeutic radioisotopes; radioactive iodine
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DA intervention (Experimental): Decision aid exposure + usual care
  Interventions: Other: Decision aid exposure
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: Decision aid exposure — Exposure to a computerized decision aid on adjuvant radioactive iodine treatment decision-making. The exposure is during one visit.
  Arms: DA intervention

SUMMARY:
In this study, we will test, using a randomized controlled trial design, whether the use of a computer-based decision aid (DA) may improve general knowledge and reduce personal decisional conflict in patients with early stage papillary thyroid cancer (PTC), when compared to usual care. Patients with early stage PTC will be required to have surgical pathologic criteria for which adjuvant RAI treatment may be considered optional.

DETAILED DESCRIPTION:
A. Primary research question

In patients with early stage papillary thyroid cancer, does the administration of a computerized decision aid improve the score on a test of knowledge about early stage PTC and adjuvant RAI treatment, when compared to usual care? (The knowledge score is a sum of positive responses from a total of 10 true/false questions in a self-administered questionnaire, to be administered at the study visit, Q2A).

B. Secondary research questions

1. In patients with early stage PTC, does the administration of a computerized decision aid reduce overall decisional conflict (as well as the following respective subscales - informed subscale, uncertainty subscale, and effective decision subscale), when compared to usual care? (Decisional Conflict questionnaire, DCS).
2. In patients with early stage PTC, does the administration of a computerized decision aid, improve reduce decisional regret relating to RAI decision making after the final decision has been made? (Decision Regret Questionnaire, DRQ)
3. In patients with early stage PTC, does the administration of a computerized decision aid, reduce the number of participants receiving adjuvant radioactive iodine treatment (analysis for all participants, as well as those who are not already on a waiting list for radioactive iodine treatment at the time of recruitment, respectively)?
4. Do the respective monitoring or blunting scores on the Miller Behavioral Style Scale (MBSS) correlate with the number of clicks for information performed by participants reviewing the decision aid? (subgroup analysis in the decision aid intervention group)
5. Do the respective monitoring or blunting scores on the Miller Behavioral Style Scale (MBSS) correlate with the score on a test of knowledge about early stage PTC and adjuvant RAI treatment? (Respective analyses planned for entire study population, as well as the intervention and control groups)
6. What are the main reasons why RAI treatment is selected or not selected (after the decision has been finalized), grouping descriptions according to exposure or non-exposure to a computerized decision aid? (See Follow-up questionnaire [administered by telephone], question 2, qualitative description, with reasons to be coded and quantified using mixed methods).

NOTE: In the original design of this study, we hoped to utilize a modified Client Satisfaction Questionnaire for assessment of satisfaction of patient participants and physicians as secondary trial outcomes. However, we are unable to utilize any modified Client Satisfaction Questionnaires in this study, because of lack of permission from the original developer of the Client Satisfaction Questionnaire-8, who has copyrighted and trademarked the questionnaire and prohibits such modifications. No modified client satisfaction questionnaire results have been analyzed in this study and will not be analyzed.

Study design The project design will be a single-centre randomized controlled trial conducted at University Health Network. The participants will be randomized to a) the decision aid group (in addition to usual care [counseling by his or her physician, called usual care]) or b) usual care. The DA will be available only to participants during the study (not the public or treating physicians). The decision aid testing will be performed at the Toronto General Hospital.

15-23 Month Extended Follow-up Study: After initiation of the primary study above, we were subsequently awarded funding to contact the enrolled study participants about 15 and 23 months post-randomization to inquire for permission to participate in an extended follow-up study. The extended follow-up study was approved by the University Health Network Research Ethics Board. Participants from the original randomized controlled trial (above) are contacted by telephone for consent to participate in the extended follow-up study, which is considered exploratory (secondary).

The extended follow-up study includes a quantitative questionnaire telephone interview component and a qualitative component. For the quantitative questionnaire component, a single telephone interview is performed updating demographics, thyroid cancer outcomes/treatments (with confirmatory medical record review and administering quantitative questionnaires verbally. A participants consenting to the extended follow-up study are also offered the opportunity to participate in an in-depth qualitative study, involving a one-on in-person interview (which is audio-recorded, transcribed, and analyzed using qualitative methods). A representative subgroup of about 15-30 participants are invited in the qualitative interview and sampling continued until saturation of themes is achieved.

The following exploratory questions are to be addressed in the quantitative component of the extended follow-up study (about 15-23 months post-randomization):

1. To what degree do participants in the study (decision aid and control groups) perceive themselves to be respectively informed and satisfied with the original radioactive iodine treatment decision? The results in respective study arms are compared.
2. To what degree do participants in the study (decision aid and control groups) perceive themselves to regret their original radioactive iodine treatment decision? The results in respective study arms are compared.
3. To what degree do participants in the study (decision aid and control groups) perceive current cancer-related worry (Assessment of Survivor Concerns Questionnaires)? The results in respective study arms are compared.
4. To what degree do participants in the study (decision aid and control groups) perceive trust in their treating physician (Trust in Physician Scale)? The results in respective study arms are compared.
5. How do participants in the study (decision aid and control groups) perceive their mood (PHQ-4 questionnaire)? The results in respective study arms are compared.

The qualitative subgroup study includes semi-structured questions on the experiences of radioactive iodine treatment decision-making, overall thyroid cancer treatment satisfaction, and study participation.

Exploratory Telephone Survey Study - 24 months or longer after randomization:

After initiation of the primary study above, we were subsequently awarded pilot study funding to contact the study participants on one occasion, two or more years post-randomization to inquire for permission to participate in an exploratory telephone survey study, intended to guide future research directions, and generate data for possible use in sample size calculations for potential future studies. The 24 month or longer post-randomization exploratory telephone survey study was approved by the University Health Network Research Ethics Board. Participants from the original randomized controlled trial (above) are contacted by telephone for consent to participate in the study, which is considered exploratory (secondary) and is thus, hypothesis-generating.

The telephone survey exploratory study (2 or more years post-randomization) consists of quantitative telephone questionnaires. A single telephone interview is performed updating demographics, thyroid cancer outcomes/treatments (with confirmatory medical record review and administering quantitative questionnaires verbally.

The following exploratory questions are to be addressed in the exploratory 24 month (or longer) post-randomization study. For all of the analyses below, descriptive data will be described for the entire study population, and if sample size permits, subgroup analyses according to decision aid status, radioactive iodine status, and age (<45 years at time of original surgery or 45 years or older at time of original surgery), and recurrence status, will be considered.

1. To describe the Cancer Impact in consenting participants, 2 or more years post-randomization. For participants in whom a negative financial impact of cancer is reported, an additional question is posed requesting explanation of this impact.
2. To describe the Information Needs of consenting participants, 2 or more years post-randomization.
3. To describe the General Concerns of consenting participants, 2 or more years post-randomization.
4. To describe cancer-related worry (Assessment of Survivor Concerns Questionnaires) two or more years following randomization.

ELIGIBILITY:
Inclusion Criteria for patient participants:

* Individuals with papillary thyroid carcinoma who have had complete resection of their thyroid at surgery (total or near-total thyroidectomy, or hemi- [subtotal] with completion thyroidectomy)on or after September 1, 2009
* Age at time of first thyroid cancer surgery must be at least 18 years or older
* The papillary thyroid cancer TNM pathologic stage must be pT1 or pT2, N0 (or Nx), M0 (or Mx) (TNM stage, AJCC VI) (ie. primary tumor size 1-4 cm, no known positive lymph nodes at the time of primary surgery, no extension of the tumor outside the thyroid, no venous or lymphatic invasion, and no known distant metastases at primary surgery, with no tall cell features, as per surgical pathology report)
* Must be able to communicate in spoken and written English
* Must be able to use a computer
* Must be able to provide informed consent on one's own (without any need for translation)

Exclusion criteria for patient participants:

* Participants not meeting inclusion criteria
* Concurrent diagnosis of medullary or anaplastic or poorly differentiated thyroid cancer or thyroid lymphoma
* Prior radioactive treatment for thyroid cancer
* Individuals who have been taken off their thyroid hormone for testing or treatment, will not be eligible for the study while off this medication.
* Individuals who are unwilling for investigators to confirm their pathologic stage of disease through review of pathology report(s) will be ineligible for the study

Inclusion criteria for the physician feedback component of this study:

- Physicians and surgeons caring for thyroid cancer patients, in active practice at University Health Network in Toronto, Ontario, Canada.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Knowledge about papillary thyroid cancer and radioactive iodine treatment | Day 0
  The knowledge questionnaire will be administered on the same day as the randomization visit (after the exposure to the decision aid for participants in the intervention group, or without exposure to the decision aid in the control group).

SECONDARY OUTCOMES:
Decisional conflict (and subscale measures) | Day 0
  The decisional conflict questionnaire will be administered on the same day as the randomization visit (after the exposure to the decision aid for participants in the intervention group, or without exposure to the decision aid in the control group).
Decisional regret | 6-12 months and 15-23 months
  Decisional regret will be assessed at least 6 months after the randomization, or later if the decision is not finalized at 6 months. The time frame should generally be about 6 - 12 months after the randomization visit. This outcome will also be evaluated at an extended follow-up study call at about 15-23 months
Reasons for accepting or declining radioactive iodine treatment | 6 - 12 months
  Rationale for accepting or declining radioactive iodine treatment will be assessed 6 months after the randomization visit as well as after the decision on radioactive iodine has been finalized (generally decision should have been finalized within 12 months).
The final decision to accept or decline adjuvant radioactive iodine treatment | 6-12 months
  The final decision to accept or decline adjuvant radioactive iodine treatment will be assessed 6 months after the randomization visit as well as after the decision on radioactive iodine has been finalized (generally decision should have been finalized within 12 months).
Feeling informed about RAI treatment decision | 15-23 months
  Questionnaire on feeling informed about a medical decision
Feeling satisfied with RAI treatment decision | 15-23 months
  Question on RAI decision satisfaction
Cancer-related worry | 15-23 months
  Assessment of Survivor Concerns questionnaire
Trust in the treating physician | 15-23 months
  Trust in Physician questionnaire
Mood | 15-23 months
  Depression and Anxiety Screen (PHQ-4) questionnaire
Qualitative data | 15-23 months
  In-depth interview, discussing RAI treatment decision-making, treatment satisfaction, and trial participation
Cancer Impact | 24 months or longer-post randomization
  Cancer Impact Questionnaire
Information Needs | 24 months or longer-post randomization
  Information Needs Questionnaire
General Concerns | 24 months or longer post-randomization
  General Concerns Questionnaire
Cancer-related Worry | 24 months or longer post-randomization
  Assessment of Survivor Concerns

CONTACTS AND LOCATIONS:
Overall Officials: Annie M Sawka, MD, PhD, Principal Investigator — University Health Network, Toronto; David P Goldstein, MD, Study Director — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Background] Sawka AM, Straus S, Brierley JD, Tsang RW, Rotstein L, Rodin G, Gafni A, Ezzat S, Thabane L, Thorpe KE, Goldstein DP. Decision aid on radioactive iodine treatment for early stage papillary thyroid cancer--a randomized controlled trial. Trials. 2010 Jul 26;11:81. doi: 10.1186/1745-6215-11-81. PMID 20659341
- [Background] Sawka AM, Straus S, Rodin G, Thorpe KE, Ezzat S, Gafni A, Goldstein DP. Decision aid on radioactive iodine treatment for early stage papillary thyroid cancer: update to study protocol with follow-up extension. Trials. 2015 Jul 14;16:302. doi: 10.1186/s13063-015-0819-6. PMID 26169592
- [Result] Sawka AM, Straus S, Rotstein L, Brierley JD, Tsang RW, Asa S, Segal P, Kelly C, Zahedi A, Freeman J, Solomon P, Anderson J, Thorpe KE, Gafni A, Rodin G, Goldstein DP. Randomized controlled trial of a computerized decision aid on adjuvant radioactive iodine treatment for patients with early-stage papillary thyroid cancer. J Clin Oncol. 2012 Aug 10;30(23):2906-11. doi: 10.1200/JCO.2011.41.2734. Epub 2012 Jul 2. PMID 22753906
- [Result] Sawka AM, Rilkoff H, Tsang RW, Brierley JD, Rotstein L, Ezzat S, Asa SL, Segal P, Kelly C, Zahedi A, Gafni A, Goldstein DP. The rationale of patients with early-stage papillary thyroid cancer for accepting or rejecting radioactive iodine remnant ablation. Thyroid. 2013 Feb;23(2):246-7. doi: 10.1089/thy.2012.0422. No abstract available. PMID 23009127
- [Result] Sawka AM, Straus S, Rodin G, Heus L, Brierley JD, Tsang RW, Rotstein L, Ezzat S, Segal P, Gafni A, Thorpe KE, Goldstein DP. Thyroid cancer patient perceptions of radioactive iodine treatment choice: Follow-up from a decision-aid randomized trial. Cancer. 2015 Oct 15;121(20):3717-26. doi: 10.1002/cncr.29548. Epub 2015 Jul 20. PMID 26195199
- [Result] Sawka AM, Straus S, Rodin G, Tsang RW, Brierley JD, Rotstein L, Segal P, Gafni A, Ezzat S, Goldstein DP. Exploring the relationship between patients' information preference style and knowledge acquisition process in a computerized patient decision aid randomized controlled trial. BMC Med Inform Decis Mak. 2015 Jun 19;15:48. doi: 10.1186/s12911-015-0168-0. PMID 26088605